CLINICAL TRIAL: NCT01107808
Title: Calcium, Vitamin D and Metformin to Treat Insulin Resistance in Obese African American Adolescent Females.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment to the study
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Stephenie Wallace, MD, UAB Department of Pedicatrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAB MHRC SBW; F090213004 (Other: UAB IRB)
Record Dates: First submitted 2010-04-01; First posted 2010-04-21 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Insulin Resistance; Insulin Sensitivity; Obesity; Vitamin D Deficiency
Keywords: Adolescents; African American; Female
MeSH Terms: conditions — Insulin Resistance; Obesity; Vitamin D Deficiency | interventions — Calcium; Ergocalciferols; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): The adolescents randomized to Standard of care group will receive the medical and behavioral counseling regarding their obesity as a patient of the Children's Center for Weight Management (CCWM). They will not receive any pharmacological treatment for their vitamin D deficiency or insulin resistance. Calcium and vitamin D dietary intake will be determined using a specific food frequency questionnaire at each study visit for all groups. This will be used to determine effect of nutrition counseling.
- Calcium and Vit D (Experimental): The participants in the vitamin D/calcium group will receive standard of care through the CCWM along with the addition of treatment with ergocalciferol (vitamin D2) and calcium carbonate for their vitamin D deficiency. The vitamin D treatment will be 50,000 IU orally weekly for 8 weeks. This treatment regimen for vitamin D deficiency has been found to be safe to children and adolescents. 32 33The dose of calcium supplementation will be calcium carbonate orally 1200mg daily. This is the daily recommended intake of calcium for adolescents
  Interventions: Drug: Calcium and Vit D
- Metformin/ Vit D (Experimental): The participants randomized into the vitamin D/calcium/Metformin treatment group will receive standard of care through the CCWM in addition to treatment for their Vitamin D deficiency with the same doses of ergocalciferol (vitamin D2) and calcium carbonate as previously outlined. Additionally, these participants will receive Metformin ER to treat insulin resistance. The Metformin ER will be started at 1000mg daily with dinner for 7 days and then increased to a final dose of 2000mg orally, daily for the remainder of the study (7 weeks).
  Interventions: Drug: Metformin, Vit D and Calcium

INTERVENTIONS:
Drug: Calcium and Vit D — ergocalciferol (vitamin D2) treatment 50,000 IU orally, weekly for 8 weeks calcium carbonate orally 1200mg daily
  Other Names: Vitamin D2 =ergocalciferol
  Arms: Calcium and Vit D
Drug: Metformin, Vit D and Calcium — ergocalciferol (vitamin D2)50,000 IU orally weekly for 8 weeks calcium carbonate orally 1200mg daily Metformin ER 1000mg daily with dinner for 7 days and then increased to a final dose of 2000mg orally, daily for the remainder of the study (7 weeks)
  Other Names: Gluophage
  Arms: Metformin/ Vit D

SUMMARY:
This is a feasibility study to examine the treatment with Metformin, vitamin D with calcium supplement for insulin resistance in obese, black, female teens. The association of low vitamin D levels and decreased insulin sensitivity has been established. Thus, the specific aims of this study are:

Specific aim 1: To examine the effect of an 8-week treatment with vitamin D and calcium supplementations on diabetes-related risk factors in obese, black, female teens.

Hypothesis 1a: In obese, black, female teens with both insulin resistance and vitamin D deficiency, treatment with vitamin D and calcium supplementation will significantly improve measures of insulin resistance and sensitivity (as determined by the homeostatic model assessment for insulin resistance and whole body insulin sensitivity index measures) when compared to controls not receiving vitamin D and calcium.

Hypothesis 1b: In obese, black teen females with both insulin resistance and vitamin D deficiency, treatment with vitamin D and calcium supplementation will significantly improve measures of cardiovascular disease (decreased BMI and improved triglycerides and LDL) when compared to controls not receiving vitamin D and calcium.

Specific aim 2: To determine if the addition of Metformin to the 8-week treatment with vitamin D and calcium supplementations improves diabetes-related risk factors in obese, black, female teens.

Hypothesis 2a: In obese, black, female teens with both insulin resistance and vitamin D deficiency, treatment with Metformin, vitamin D, and calcium supplementation will significantly improve measures of insulin resistance and sensitivity (as determined by the homeostatic model assessment for insulin resistance and whole body insulin sensitivity index measures) when compared to standard of care or treatment with vitamin D with calcium supplementation alone while controlling for dietary intake of vitamin D and calcium.

Hypothesis 2b: In obese, black, female teens with both insulin resistance and vitamin D deficiency, treatment with Metformin, vitamin D, and calcium supplementation will significantly improve measures of cardiovascular disease risk (as determined by the decreased BMI, improved triglycerides and LDL) when compared to standard of care or treatment with vitamin D with calcium supplementation alone while controlling for dietary intake of vitamin D and calcium.

DETAILED DESCRIPTION:
The increasing rate of obesity in youth has reached epidemic proportion in the United States. African Americans share an overwhelming burden of this disorder and its complications.1 Vitamin D deficiency is prevalent in black girls and women2 and is associated with insulin resistance in populations at risk for diabetes.3 The use of Metformin, an oral diabetic agent, to halt the progression to diabetes in individuals at risk has been studied, but not in a population with concurrent vitamin D deficiency. In this proposal, we hypothesize that treatment with vitamin D with calcium supplement along with Metformin together will improve insulin resistance in obese, black teen girls. We will investigate this hypothesis in two specific aims to: 1) examine the effect of treatment of Vitamin D deficiency on insulin resistance in mature black teen girls, 2) to determine if there is any additional benefit of Metformin with treatment for Vitamin D deficiency to improve insulin resistance in this group. We propose to accomplish these aims through a clinical trial in obese black teen girls who have reached developmental maturity (approximately 15-18 years old) with vitamin D deficiency. Eligible participants will be randomized to one of three groups: standard of care, treatment with vitamin D/calcium supplement, and treatment with Vitamin D/Calcium Supplement and Metformin. We will enroll 30 obese adolescent subjects, (10 participants per group) into this 2-month study. The following measurements will be performed at baseline and 2 month follow-up: a) 25-hydroxy-vitamin D, b) Oral glucose tolerance tests to calculate homeostatic model assessment for insulin resistance (HOMA IR), and 4 to determine insulin resistance and total body insulin sensitivity index (TBISI) to determine insulin sensitivity,5 c) body mass index calculations, and c) lipid panel to include triglyceride, HDL-C, and LDL-C measurements. We will control for the effect of nutritional counseling on vitamin D and calcium intake will be controlled. Our outcome measures will include improvement in insulin resistance and decreased body mass index for our participants treated with vitamin D, calcium supplementation and Metformin. Validation of our hypothesis will show that Metformin along with vitamin D treatment and calcium supplementation is a novel treatment combination to improve insulin resistance, the health of an at-risk adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* 14-19 years old
* female
* african american
* obese
* risk of insulin resistance (physical exam or family history of diabetes
* willing to be randomized to a arm that would take medication

Exclusion Criteria:

* pregnancy
* male
* kidney or liver dysfunction
* unwilling to take pill/medication during the trial interested in becoming pregnant

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-09 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
The insulin sensitivity indices (HOMA IR) | 8 weeks
  the HOMA IR will be calculated from glucose and insulin measurements from the OGTT done at the screening and final study visits.

SECONDARY OUTCOMES:
Low-density lipoprotein LDL | 8 week
  LDL-C will be measured by standard laboratory methods through the hospital clinic lab.The screening and final measurement will be compared for each participant.
The insulin sensitivity indices (WBISI) | 8 weeks
  the WBISI will be calculated from glucose and insulin measurements from the OGTT done at the screening and final study visits.
High density lipoprotein | 8 weeks
  HDL will be measured by standard laboratory methods through the hospital clinic lab. The screening and final measurement will be compared for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Stephenie B Wallace, Principal Investigator — UAB Department of Pediatrics